CLINICAL TRIAL: NCT02121808
Title: Evaluation of Different Pre-Oxygenation Conditions in Morbid Obesity: Position and Ventilation Mode, in a Respiratory Physiology Laboratory, on Voluntary Subjects
Brief Title: EPO2-PV: Evaluation of Pre-Oxygenation Conditions in Morbidly Obese Volunteer: Effect of Position and Ventilation Mode
Acronym: EPO2-PV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean Bussières, Anesthesiologist, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IUCPQ 21054
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2017-09

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate
Keywords: Morbid Obesity; Bariatric Surgery Candidate; Pre-Oxygenation; Functional Residual Capacity
MeSH Terms: conditions — Obesity, Morbid | interventions — Tidal Volume

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Supine (Experimental): NIPPV and Tidal volume
  Interventions: Procedure: NIPPV; Procedure: Tidal volume
- Beach-chair (Back : 25 deg) (Experimental): NIPPV and Tidal volume
  Interventions: Procedure: NIPPV; Procedure: Tidal volume
- Proclive (Global 25 deg) (Experimental): NIPPV and Tidal volume
  Interventions: Procedure: NIPPV; Procedure: Tidal volume

INTERVENTIONS:
Procedure: NIPPV — Ventilation: non-invasive positive pressure ventilation (NIPPV)
  Positive end-expiratory pressure: 10 cmH20 Pressure support: 5 - 20 cm H2O for tidal volume of 10 mL / kg (ideal body weight)
Procedure: Tidal volume — Tidal volume spontaneous ventilation, no assistance.

SUMMARY:
The risk of complications associated with airway management in obese patients is significant. The results of pre-oxygenation allow a prolonged non-hypoxic apnea time for the clinician. The increase in FRC and non-hypoxic apnea time is correlated. The best condition to accomplish the pre-oxygenation in morbidly obese patient is still undetermined in medical literature.

This study is designed to evaluate the effect of different positions combined with different ventilation modes during the pre-oxygenation phase of anesthesia's induction. EPO2: PV will evaluate the effect of different combinations of positions and ventilation modes on pulmonary volumes (mainly functional residual capacity) in a morbidly obese volunteer.

DETAILED DESCRIPTION:
Complications related to airway management are the major contributing factor to morbidity in anesthesiology. This risk of complications markedly increases when faced with a difficult airway in an obese patient. Pre-oxygenation creates a safety margin by increasing the patient's oxygen stores, through a higher functional residual capacity (FRC). When pre-oxygenated, the clinician may proceed to intubation after a variable period of apnea, while maintaining oxygen saturation over 92%. In non-obese individuals, pre-oxygenation allows a non-hypoxic apnea time of eight minutes. In the obese population, however, this non-hypoxic apnea time decreases to two to three minutes.

Different methods of pre-oxygenation have been proposed in order to increase apnea time before significant oxygen desaturation. Amongst these methods, the following are of particular interest: pre-oxygenation to vital capacity, pre-oxygenation with spontaneous ventilation and positive pressure, and pre-oxygenation with elevated head positioning ("beach-chair"). These methods have been extensively studied in individuals of normal height and weight.

The main objective of pre-oxygenation is to raise oxygen levels available at the alveolar level in order to increase the non-hypoxic apnea time, before a significant desaturation occurs. This raised alveolar oxygen concentration can be done by maintaining a higher inspired oxygen fraction and by promoting a larger FRC which is the oxygen reserve build through the pre-oxygenation phase. In morbid obese patients, these parameters are affected by a lower expiratory flow, lower expiratory flow and closing of small radius airways. The final result probably come from a more cephalad position of the diaphragm induced by a larger intra-abdominal volume.

Actually, different studies demonstrate the advantage of a beach-chair position and non-invasive positive pressure ventilation for pre-oxygenation of obese patients. These advantages are shown by a shorter time of pre-oxygenation to obtain an end-tidal O2 > 90 % and a longer non-hypoxic apnea time (Sat O2 >90%). Up to date, there is no published data on the FRC as a result of different combinations of position and ventilation mode. This study will evaluate FRC by helium dilution technique.

We propose a crossover randomised trial on volunteers waiting for a bariatric surgery. We want to compare, in pre-oxygenation situation, without induction of general anesthesia, the effect of three positions and two ventilation modes on the FRC measure.

ELIGIBILITY:
Inclusion Criteria:

* BMI 40 - 80 kg / m2
* Waist circumference: Men: More than 130 cm
* Waist circumference: Women: More than 115 cm

Exclusion Criteria:

* Facial hair
* Cranio-facial abnormality
* Claustrophobia
* Asthma
* COPD (defined by FEV1 < 80 %)
* Severe cardiovascular disease (defined by NYHA ≥3)
* Pregnancy
* Tobacco use
* NI-CPPV Intolerance documented by a respiratory specialist (pneumologist).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne J Couture, MD, Principal Investigator — Laval University; Jean S Bussières, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Cheney FW, Posner KL, Lee LA, Caplan RA, Domino KB. Trends in anesthesia-related death and brain damage: A closed claims analysis. Anesthesiology. 2006 Dec;105(6):1081-6. doi: 10.1097/00000542-200612000-00007. PMID 17122570
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Juvin P, Lavaut E, Dupont H, Lefevre P, Demetriou M, Dumoulin JL, Desmonts JM. Difficult tracheal intubation is more common in obese than in lean patients. Anesth Analg. 2003 Aug;97(2):595-600. doi: 10.1213/01.ANE.0000072547.75928.B0. PMID 12873960
- [Background] Campbell IT, Beatty PC. Monitoring preoxygenation. Br J Anaesth. 1994 Jan;72(1):3-4. doi: 10.1093/bja/72.1.3. No abstract available. PMID 8110546
- [Background] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Background] Benumof JL, Dagg R, Benumof R. Critical hemoglobin desaturation will occur before return to an unparalyzed state following 1 mg/kg intravenous succinylcholine. Anesthesiology. 1997 Oct;87(4):979-82. doi: 10.1097/00000542-199710000-00034. No abstract available. PMID 9357902
- [Background] Berthoud MC, Peacock JE, Reilly CS. Effectiveness of preoxygenation in morbidly obese patients. Br J Anaesth. 1991 Oct;67(4):464-6. doi: 10.1093/bja/67.4.464. PMID 1931404
- [Background] Murphy C, Wong DT. Airway management and oxygenation in obese patients. Can J Anaesth. 2013 Sep;60(9):929-45. doi: 10.1007/s12630-013-9991-x. Epub 2013 Jul 9. PMID 23836064
- [Background] Tanoubi I, Drolet P, Donati F. Optimizing preoxygenation in adults. Can J Anaesth. 2009 Jun;56(6):449-66. doi: 10.1007/s12630-009-9084-z. Epub 2009 Apr 28. PMID 19399574
- [Background] Parameswaran K, Todd DC, Soth M. Altered respiratory physiology in obesity. Can Respir J. 2006 May-Jun;13(4):203-10. doi: 10.1155/2006/834786. PMID 16779465
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Boyce JR, Ness T, Castroman P, Gleysteen JJ. A preliminary study of the optimal anesthesia positioning for the morbidly obese patient. Obes Surg. 2003 Feb;13(1):4-9. doi: 10.1381/096089203321136511. PMID 12630606
- [Background] Burns SM, Egloff MB, Ryan B, Carpenter R, Burns JE. Effect of body position on spontaneous respiratory rate and tidal volume in patients with obesity, abdominal distension and ascites. Am J Crit Care. 1994 Mar;3(2):102-6. PMID 8167771
- [Background] Coussa M, Proietti S, Schnyder P, Frascarolo P, Suter M, Spahn DR, Magnusson L. Prevention of atelectasis formation during the induction of general anesthesia in morbidly obese patients. Anesth Analg. 2004 May;98(5):1491-5, table of contents. doi: 10.1213/01.ane.0000111743.61132.99. PMID 15105237
- [Background] Gander S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Positive end-expiratory pressure during induction of general anesthesia increases duration of nonhypoxic apnea in morbidly obese patients. Anesth Analg. 2005 Feb;100(2):580-584. doi: 10.1213/01.ANE.0000143339.40385.1B. PMID 15673897
- [Background] Delay JM, Sebbane M, Jung B, Nocca D, Verzilli D, Pouzeratte Y, Kamel ME, Fabre JM, Eledjam JJ, Jaber S. The effectiveness of noninvasive positive pressure ventilation to enhance preoxygenation in morbidly obese patients: a randomized controlled study. Anesth Analg. 2008 Nov;107(5):1707-13. doi: 10.1213/ane.0b013e318183909b. PMID 18931236
- [Background] Futier E, Constantin JM, Pelosi P, Chanques G, Massone A, Petit A, Kwiatkowski F, Bazin JE, Jaber S. Noninvasive ventilation and alveolar recruitment maneuver improve respiratory function during and after intubation of morbidly obese patients: a randomized controlled study. Anesthesiology. 2011 Jun;114(6):1354-63. doi: 10.1097/ALN.0b013e31821811ba. PMID 21478734
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Derived] Couture EJ, Provencher S, Somma J, Lellouche F, Marceau S, Bussieres JS. Effect of position and positive pressure ventilation on functional residual capacity in morbidly obese patients: a randomized trial. Can J Anaesth. 2018 May;65(5):522-528. doi: 10.1007/s12630-018-1050-1. Epub 2018 Jan 18. PMID 29435810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was held between April 14th 2014 and June 26th 2014 by telephonic solicitation and through the preoperative bariatric clinic of our institution.
Groups:
- Position and Spontaneous vs Pressure Support: The effect of position and spontaneous vs pressure support ventilation on FRC was assessed on patients recruited. The six possible combination were tested on every patients in a randomized order.
  Intervention 1 : Supine + NIPPV Intervention 2 : Supine + Tidal volume spontaneous ventilation Intervention 3 : Beach chair (Back 25 deg) + NIPPV Intervention 4 : Beach chair (Back 25 deg) + Tidal volume spontaneous ventilation Intervention 5 : Proclive (Global 25 deg) + NIPPV Intervention 6 : Proclive (Global 25 deg) + Tidal volume spontaneous ventilation
Period: Overall Study
Arm/Group | Position and Spontaneous vs Pressure Support
Started | 20
Completed | 17
Not Completed | 3
Not completed — Technical problem | 3

BASELINE CHARACTERISTICS:
Arm/Group | Position and Spontaneous vs Pressure Support
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 5
BMI [Mean (Standard Deviation); unit: kg/m2] | 50 (8)
Waist circumference [Mean (Standard Deviation); unit: cm] | 143 (17)

OUTCOME MEASURES:

1. Primary Outcome: Functional Residual Capacity
Description: Change of functional residual capacity (FRC), in obese patient, as a result of different pre-oxygenation positions; 1- supine, 2-beach-chair, 3- reverse Trendelenburg, in two different ventilation modes : 1- spontaneous ventilation at tidal volume, 2- non-invasive positive pressure ventilation with inspiratory assistance.
Time Frame: After a 5 minutes pre-oxygenation period
Measure: Mean (Standard Deviation); unit: ml
Groups:
- 1. Supine + NIPPV: Intervention 1 : Supine + NIPPV
- 2. Supine + Tidal Volume Spontaneous Ventilation: Intervention 2 : Supine + Tidal volume spontaneous ventilation
- 3. Beach Chair (Back 25 Deg) + NIPPV: Intervention 3 : Beach chair (Back 25 deg) + NIPPV
- 4. Beach Chair (Back 25 Deg) + Tidal Volume Spontaneous Ventil: Intervention 4 : Beach chair (Back 25 deg) + Tidal volume spontaneous ventilation
- 5. Proclive (Global 25 Deg) + NIPPV: Intervention 5 : Proclive (Global 25 deg) + NIPPV
- 6. Proclive (Global 25 Deg) + Tidal Volume Spontaneous Ventila: Intervention 6 : Proclive (Global 25 deg) + Tidal volume spontaneous ventilation
Arm/Group | 1. Supine + NIPPV | 2. Supine + Tidal Volume Spontaneous Ventilation | 3. Beach Chair (Back 25 Deg) + NIPPV | 4. Beach Chair (Back 25 Deg) + Tidal Volume Spontaneous Ventil | 5. Proclive (Global 25 Deg) + NIPPV | 6. Proclive (Global 25 Deg) + Tidal Volume Spontaneous Ventila
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
ml | 2573 (515) | 2145 (438) | 2456 (442) | 2219 (477) | 2684 (473) | 2282 (501)

2. Secondary Outcome: Diaphragmatic Amplitude.
Description: Evaluation of changes in diaphragmatic amplitude and movement determined by fluoroscopy imaging after a 5 minutes pre-oxygenation period in the 6 combinations previously described.
Time Frame: After a 5 minutes pre-oxygenation period
Reporting Status: Not Posted

3. Secondary Outcome: Respiratory Mechanics
Description: Change in respiratory mechanics (compliance, resistance, tidal volume, positive end-expiratory pressure, maximal inspiratory pressure) evaluated at the end of a 5 minutes pre-oxygenation period in the 6 combinations previously described.
Time Frame: At the end of a 5 minutes pre-oxygenation period
Reporting Status: Not Posted

4. Secondary Outcome: Patient's Comfort
Description: Evaluation of the patient's comfort at the end of each intervention on an analog visual scale after a 5 minutes pre-oxygenation period in the 6 combinations previously described.
Time Frame: At the end of a 5 minutes pre-oxygenation period
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Vital Signs
Description: Change in vital signs before and after the pre-oxygenation phase in the 6 combinations after a 5 minutes pre-oxygenation period in the 6 combinations previously described.
Time Frame: At the end of a 5 minutes pre-oxygenation period
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Position and Spontaneous vs Pressure Support
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No